CLINICAL TRIAL: NCT06793059
Title: Evaluation of Flow Diverter Technology Device for Intracranial Aneurysm (SHIELD)
Acronym: SHIELD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carlos Pena, PhD, MS (Other)
Responsible Party: Sponsor-Investigator, Carlos Pena, PhD, MS, Chief Regulatory Officer, Jacobs institute
Organization: Jacobs institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001; SHIELD (Other: Jacobs Institute)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SHIELD Study Arm (Other): Active treatment with the Pipeline SHIELD Device
  Interventions: Device: SHIELD

INTERVENTIONS:
Device: SHIELD — Pipeline SHIELD device under study

SUMMARY:
The Jacobs Institute is participating in a study designed to collect prospective clinical evidence to evaluate the approved use of the Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with wide-necked intracranial aneurysms

DETAILED DESCRIPTION:
The Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments. The Pipeline™ Flex Embolization Device with Shield Technology™ is also indicated for use in the internal carotid artery up to the terminus for the endovascular treatment of adults (22 years of age or older) with small and medium wide-necked (neck width ≥ 4 mm or dome-to-neck ratio < 2) saccular or fusiform intracranial aneurysm (IAs) arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* Adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments.

Exclusion Criteria:

Exclusion Criteria:

* Cannot provide consent or legally authorized representative not available to provide consent Criteria:

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of thromboembolic event(s) | 12 Months
  The Pipeline™ Flex Embolization Device with Shield Technology™ for the endovascular treatment of adults (22 years of age or older) with large or giant wide-necked intracranial aneurysms (IAs) in the internal carotid artery from the petrous to the superior hypophyseal segments. The Pipeline™ Flex Embolization Device with Shield Technology™ is also indicated for use in the internal carotid artery up to the terminus for the endovascular treatment of adults (22 years of age or older) with small and medium wide-necked (neck width ≥ 4 mm or dome-to-neck ratio < 2) saccular or fusiform intracranial aneurysm (IAs) arising from a parent vessel with a diameter ≥ 2.0 mm and ≤ 5.0 mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobs Institute, Buffalo, New York, United States